CLINICAL TRIAL: NCT01234207
Title: Clinical Assessment of a Customized Free-form Progressive Addition Lens Spectacle
Acronym: CZV_PAL1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: Carl Zeiss Meditec, Inc. (Industry)
Responsible Party: Principal Investigator, Meng C. Lin, Director, Clinical Research Center, University of California, Berkeley
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CZV_PAL1
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Presbyopia
Keywords: Progressive addition lenses; Customized free-form; Presbyopia; Bifocals; Subjective assessment; Visual performance; Visual acuity; Amsler grid
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Randomized Order of Interventions 1 (Active Comparator): Randomized to first wear standard, non-free-form, non-customized PAL spectacles, then second, crossover to wear individually customized free-form surfaced PAL spectacles
  Interventions: Device: Standard, non-free-form, non-customized PAL spectacles; Device: Individually customized free-form surfaced PAL spectacles
- Randomized Order of Interventions 2 (Active Comparator): Randomized to first wear individually customized free-form surfaced PAL spectacles, then second, crossover to wear standard, non-free-form, non-customized PAL spectacles
  Interventions: Device: Standard, non-free-form, non-customized PAL spectacles; Device: Individually customized free-form surfaced PAL spectacles

INTERVENTIONS:
Device: Standard, non-free-form, non-customized PAL spectacles — Control spectacles include several different PAL brands as selected by patients in the UC Berkeley Optometry Clinic and purchased in the Eyewear Center; after successful fitting and purchase, potential subjects were recruited for the trial.
Device: Individually customized free-form surfaced PAL spectacles — Test spectacles are Zeiss Individual, free-form surfaced, and customized using the iTerminal device to account for individual back vertex distance, wrap angle and pantoscopic tilt
  Other Names: Zeiss Individual, Carl Zeiss Vision, Inc., Germany

SUMMARY:
The purpose of this study was to compare objective clinical measures of visual performance and subjective measures of satisfaction and preference between standard progressive addition lens (PAL) spectacles and a new type of free-form surfaced, optically customized PAL spectacle.

DETAILED DESCRIPTION:
In a double-masked crossover trial, 95 experienced wearers wore customized free-form PAL spectacles (Test) and standard non-free-form PAL spectacles (Control) for one week each. All subjects wore both Test and Control spectacles, and the pair to be worn first was randomly assigned. At dispensing and after 1 week of wear, subjects were tested for distance and near visual acuity (VA) under both high and low contrast; in addition, 30 degree off-axis VA was measured using a novel apparatus, as was the horizontal extent of undistorted vision at reading distance. Subjects also completed a set of questionnaires detailing their satisfaction levels, adaptation times, and preferences for Test or Control spectacles for different visual tasks.

ELIGIBILITY:
Inclusion Criteria:

* Presbyope
* Experienced PAL spectacle wearer
* Correctable to at least 20/25 in both eyes
* Able and willing to use Test and Control spectacles for 1 week each as primary form of presbyopia correction
* Able and willing to complete all laboratory measurements and questionnaire batteries

Exclusion Criteria:

* Purchasing free-form PAL spectacles from the UC Berkeley Eyewear Center
* Having eye conditions or diseases that could potentially cause a decrease in visual acuity over the course of participation in the study
* Having eye conditions or diseases that could potentially interfere with ability to use Test and Control spectacles as primary form of presbyopia correction

Ages: 39 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2009-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meng C. Lin, OD, PhD, Principal Investigator — Clinical Research Center, School of Optometry, University of California, Berkeley
Locations (1):
- Clinical Research Center, School of Optometry, University of California, Berkeley, Berkeley, California, United States

REFERENCES:
- [Result] Han SC, Graham AD, Lin MC. Clinical assessment of a customized free-form progressive add lens spectacle. Optom Vis Sci. 2011 Feb;88(2):234-43. doi: 10.1097/OPX.0b013e31820846ac. PMID 21217408

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Presbyopic subjects were recruited from the population of patients who were purchasing non-free-form PAL spectacles with antireflective coating in new frames from the University of California, Berkeley School of Optometry Eyewear Center.
Pre-assignment Details: 95 subjects were recruited, all of whom met the eligibility criteria and completed the study.
Groups:
- Group 1 - Control Spectacles Worn First, Then Test Spectacles: Crossover trial; 2 arms: subjects randomized to wear Control spectacles 1st, then Test spectacles 2nd
- Group 2 - Test Spectacles Worn First, Then Control Spectacles: Crossover trial; 2 arms: subjects randomized to wear Test spectacles 1st, then Control spectacles 2nd
Period: First Intervention
Arm/Group | Group 1 - Control Spectacles Worn First, Then Test Spectacles | Group 2 - Test Spectacles Worn First, Then Control Spectacles
Started | 47 | 48
Completed | 47 | 48
Not Completed | 0 | 0
Period: 1-Week Washout Period
Arm/Group | Group 1 - Control Spectacles Worn First, Then Test Spectacles | Group 2 - Test Spectacles Worn First, Then Control Spectacles
Started | 47 | 48
Completed | 47 | 48
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Group 1 - Control Spectacles Worn First, Then Test Spectacles | Group 2 - Test Spectacles Worn First, Then Control Spectacles
Started | 47 | 48
Completed | 47 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Crossover trial: all study participants received both Test and Control spectacles, in randomized order.
Arm/Group | All Study Participants
Number analyzed (Participants) | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 80
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 73
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 95

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity, High Contrast, Distance Chart
Description: Standard assessment of high contrast visual acuity at distance, as in normal clinical practice, using Baily-Lovey charts and the M&S Technologies Smart System II visual acuity projection system.
Time Frame: Post-1 week of wear of Test Spectacles and post-1 week of wear of Control Spectacles
Population: 95 presbyopic subjects wearing standard, non-free-form, non-customized PAL spectacles for 1 week, and individually customized, free-form surfaced PAL spectacles for 1 week, in randomized order, with a 1-week washout period
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Control Spectacles; Test Spectacles: Arm/Groups Outcome Measures are reported "per intervention".
Arm/Group | Control Spectacles | Test Spectacles
Number analyzed (Participants) | 95 | 95
logMAR | -0.12 (0.06) | -0.11 (0.07)

2. Primary Outcome: Visual Acuity, Low Contrast, Distance Chart
Description: Standard assessment of low contrast visual acuity at distance, as in normal clinical practice, using Baily-Lovey charts and the M&S Technologies Smart System II visual acuity projection system.
Time Frame: Post-1 week of wear of Test Spectacles and post-1 week of wear of Control Spectacles
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Control Spectacles | Test Spectacles
Number analyzed (Participants) | 95 | 95
logMAR | 0.01 (0.07) | 0.01 (0.07)

3. Primary Outcome: Visual Acuity, High Contrast, Near Chart
Description: Standard assessment of high contrast visual acuity at near, as in normal clinical practice, using Baily-Lovey charts and the M&S Technologies Smart System II visual acuity projection system.
Time Frame: Post-1 week of wear of Test Spectacles and post-1 week of wear of Control Spectacles
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Control Spectacles | Test Spectacles
Number analyzed (Participants) | 95 | 95
logMAR | -0.11 (0.13) | -0.09 (0.09)

4. Primary Outcome: Visual Acuity, Low Contrast, Near Chart
Description: Standard assessment of low contrast visual acuity at near, as in normal clinical practice, using Baily-Lovey charts and the M&S Technologies Smart System II visual acuity projection system.
Time Frame: Post-1 week of wear of Test Spectacles and post-1 week of wear of Control Spectacles
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Control Spectacles | Test Spectacles
Number analyzed (Participants) | 95 | 95
logMAR | 0.05 (0.09) | 0.12 (0.64)

5. Primary Outcome: 30-degree Off-axis Distance Visual Acuity, High Contrast Chart
Description: Measured with subject immobilized in specially designed apparatus, keeping head pointed straight forward and moving only the eyes to left or right to view the off-axis chart
Time Frame: Post-1 week of wear of Test Spectacles and post-1 week of wear of Control Spectacles
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Control Spectacles | Test Spectacles
Number analyzed (Participants) | 95 | 95
logMAR
  Off-Axis Left | 0.10 (0.13) | 0.10 (0.14)
  Off-Axis Right | 0.05 (0.09) | 0.04 (0.10)

6. Primary Outcome: 30-degree Off-axis Distance Visual Acuity, Low Contrast Chart
Description: as for outcome 5
Time Frame: Post-1 week of wear of Test Spectacles and post-1 week of wear of Control Spectacles
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Control Spectacles | Test Spectacles
Number analyzed (Participants) | 95 | 95
logMAR
  Off-Axis Left | 0.24 (0.12) | 0.24 (0.12)
  Off-Axis Right | 0.19 (0.10) | 0.16 (0.11)

7. Primary Outcome: Horizontal Extent of Undistorted Vision at Reading Distance
Description: Novel apparatus designed to immobilize head and allow subject to indicate point of peripheral optical distortion on a modified Amsler-type grid
Time Frame: Post-1 week of wear of Test Spectacles and post-1 week of wear of Control Spectacles
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Control Spectacles | Test Spectacles
Number analyzed (Participants) | 95 | 95
cm | 17.74 (9.87) | 20.06 (11.89)

8. Primary Outcome: Questionnaire Battery
Description: Forced-choice Likert scale preference questionnaire
Time Frame: At study exit, after both Test and Control spectacles had been worn for 1 week each
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Control Spectacles | Test Spectacles
Number analyzed (Participants) | 95 | 95
percentage of participants
  Overall Preference | 45 | 55
  Preference for Distance Vision | 40 | 60
  Preference for Active Vision | 40 | 60
  Preference for Midrange Vision | 45 | 55
  Preference for Transitional Vision | 45 | 55
  Preference for Near Vision | 50 | 50

ADVERSE EVENTS:
Time Frame: 9 months (study duration)
Groups:
- Control Spectacles; Test Spectacles: Arm/Groups Adverse Events are reported "per intervention"
Arm/Group | Control Spectacles | Test Spectacles
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/95
Other Adverse Events (participants affected / at risk) | 0/95 | 0/95

LIMITATIONS AND CAVEATS:
Possibility of insufficient head immobilization during off-axis VA measurement on left side only for some subjects. May explain difference of off-axis VA results between right and left sides.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No